CLINICAL TRIAL: NCT02056028
Title: Validation of Our Policy of Long-term Drains Maintenance After Hepatic Resection: Results of a Prospective Cohort Analysis
Brief Title: Bile Leak After Liver Surgery
Status: Completed | Type: Observational
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Prof. Guido Torzilli, Professor of Surgery, University of Milan
Other Study IDs: BileLeakLiverSurgery
Record Dates: First submitted 2014-02-03; First posted 2014-02-05 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Bile Leak; Hepatic Resection; Liver Resection; Hepatectomy; Biliary Fistula
MeSH Terms: conditions — Biliary Fistula | interventions — Hepatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Bile leak after hepatic resection
  Interventions: Procedure: Hepatic resection

INTERVENTIONS:
Procedure: Hepatic resection
  Other Names: Liver resection; Hepatectomy

SUMMARY:
The definition of biliary fistula is heterogeneous and the more accepted is that proposed by the ISGLS. We devised a precise definition of post-resectional biliary fistula and a well-established policy both for its disclosure and management.Aim was the validation of our definition, and management of biliary fistula after hepatic resection in a large prospective cohort of patients and its comparison with that of the International Study Group of Liver Surgery (ISGLS).

DETAILED DESCRIPTION:
Data on abdominal drains and on clinical, pathological and short-term outcome were reviewed in a prospective cohort of patients who underwent hepatic resection between 2004 and 2012. Drains were maintained at least 7 days, and the bilirubin levels were measured in POD3, 5, and 7. Drains were removed if the bilirubin level in POD7 was inferior than in POD5, and less than 10 mg/dl. Statistical analysis on prognostic factors for biliary fistula was performed.

ELIGIBILITY:
Inclusion Criteria:

* any patient submitted to hepatic resection at our Unit between the established frame time

Exclusion Criteria:

* any patient with incomplete data or follow-up

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The records of 475 consecutive patients who were submitted to hepatectomy between 2004-2012 were reviewed.
Sampling Method: Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2004-01; Primary Completion 2012-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Bile leak | 7 days
  The first study endpoint was the ability of our criteria to detect and manage bile leak after liver surgery. For this purpose we considered the rate of bile leaks detected and managed using the surgical drains, and the rate of abdominal collections that required any surgical or radiological intervention after drains removal.

SECONDARY OUTCOMES:
ISGLS definition | 7 days
  The second endpoint was the exploration of the ISGLS definition of bile leak in the herein presented cohort of patients in regards of the rate of bile leaks and abdominal collections.
ISGLS definition | 90 days
  Exploration of reliability and efficacy of the International Study Group on Liver Surgery (ISGLS) definition of bile leak after hepatectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Milan, Italy

REFERENCES:
- [Background] Torzilli G, Olivari N, Del Fabbro D, Gambetti A, Leoni P, Gendarini A, Makuuchi M. Bilirubin level fluctuation in drain discharge after hepatectomies justifies long-term drain maintenance. Hepatogastroenterology. 2005 Jul-Aug;52(64):1206-10. PMID 16001662
- [Derived] Donadon M, Costa G, Cimino M, Procopio F, Del Fabbro D, Palmisano A, Torzilli G. Diagnosis and Management of Bile Leaks After Hepatectomy: Results of a Prospective Analysis of 475 Hepatectomies. World J Surg. 2016 Jan;40(1):172-81. doi: 10.1007/s00268-015-3143-0. PMID 26148518